CLINICAL TRIAL: NCT02534376
Title: Phase 0 Trial of Presurgical Cholesterol-lowering on Prostate Cancer Cell Growth
Brief Title: Cellular Effect of Cholesterol-Lowering Prior to Prostate Removal
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Principal Investigator, Hyung L. Kim, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00040945
Record Dates: First submitted 2015-08-25; First posted 2015-08-27 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: prostatectomy, cholesterol, statin
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ezetimibe; Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Vytorin (ezetimibe 10mg-simvastatin 40mg)
  Interventions: Drug: ezetimibe 10mg-simvastatin 40mg

INTERVENTIONS:
Drug: ezetimibe 10mg-simvastatin 40mg — Vytorin (ezetimibe 10mg-simvastatin 40mg) will be given on an outpatient basis. The drug will be taken orally each day until the subject undergoes radical prostatectomy. The start of Vytorin is timed so that patients get the last dose the day before surgery. Subjects receive a two to four weeks of Vytorin.
  Other Names: Vytorin

SUMMARY:
There is evidence in human studies as well as animal studies that treatments to lower cholesterol can reduce the risk of dying from prostate cancer.To decide if cholesterol-lowering therapy can slow the growth of prostate cancer, the investigators would like to lower cholesterol prior to surgery and then measure the growth of prostate cancers cells when the prostate has been removed. The investigators will use the combination of two drugs that is approved by the U.S. Food and Drug Administration to lower cholesterol. The drug combination is commercially available with a doctor's prescription and sold as Vytorin®. It is known that maximal cholesterol-lower effects are seen after 2 weeks of treatment with Vytorin®. Therefore, study patients receive at least 2 weeks, but no more than 6 weeks of Vytorin® prior to surgery.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

Prostate cancer is the most commonly diagnosed cancer and the second leading cause of cancer death among men in North America. In the US, there are more than 200,000 newly diagnosed cases and nearly 40,000 deaths from prostate cancer (CaP) annually. Although elevated lipid levels are understood to increase risk of coronary heart disease, their importance for CaP is not understood. Epidemiologic studies consistently show an association between lipid lowering interventions and decreased risk of advanced CaP. There are no reports of prospective studies of lipid-lowering interventions directed at CaP.

Epidemiologic studies and preclinical observations suggest that interventions to lower cholesterol will decrease the risk of developing lethal CaP. However, a definitive, phase III study of cholesterol-lowering effects on advanced CaP development is needed prior to clinical implementation of this intervention. Such a trial will require a massive commitment of resources for the large number of patients needing long follow-up. A rational intermediate step is to conduct a presurgical intervention study to lower cholesterol in men undergoing radical prostatectomy. Molecular evidence of treatment effect will provide a sound rationale for definitive clinical trials, and may provide predictive biomarkers that can be validated in these future trials.

The investigators propose a prospective trial to assess the effects on the human prostate of a maximal cholesterol lowering strategy using dual agents in men already scheduled to undergo radical prostatectomy for prostate cancer.

Simvastatin is a cholesterol-lowering drug approved by the FDA in 1991 and is now commercially available as Zocor (Merck) or as a generic agent. After ingestion, it is converted from an inactive lactone to the corresponding β-hydroxyacid, which inhibits HMG-CoA reductase and the conversion of HMG-CoA to mevalonate. Ezetimibe is a cholesterol-lowering agent that operates by a distinct mechanism from HMG-CoA reductase inhibitors. It was FDA approved in 2002 and is commonly administered alone or in combination with a statin. It specifically inhibits a cholesterol transporter in the small intestines and selectively inhibits the absorption of cholesterol and related sterols.

A single pill that combines simvastatin and ezetimibe is available from Merck (Vytorin). This commercially available agent at its standard dose is used in this trial. This study uses the combination of simvastatin and ezetimibe to achieve maximal cholesterol lowering prior to prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy containing ≥ 10 tissue cores sampled
* Biopsy positive for adenocarcinoma of the prostate containing any quantity of Gleason 3 component (e.g. Gleason score 3+3, 3+4, 4+3)
* Scheduled to undergo robotic radical prostatectomy
* Serum Prostate-Specific Antigen (PSA) <20 ng/ml
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Pharmacologic therapy (e.g. statins or ezetimibe) to lower cholesterol within 30 days prior to registration.
* Prior treatment for CaP by surgery, irradiation, local ablative (e.g. cryosurgery or high intensity focused ultrasound) or androgen deprivation therapy.
* 5-alpha reductase inhibitors (e.g. finasteride or dutasteride) within 180 days prior to registration.
* Hypersensitivity to simvastatin or ezetimibe.
* Pharmacologic therapy with agents reported to produce adverse drug-drug interactions. (Table 2)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Growth of Gleason grade 3 prostate cancer | following 2-6 weeks of cholesterol lowering intervention.
  Prostate tissue removed at the time of surgery will be examined to measure cellular growth using molecular assays.

SECONDARY OUTCOMES:
Growth of benign prostate glands | following 2-6 weeks of cholesterol lowering intervention.
  Prostate tissue removed at the time of surgery will be examined to measure cellular growth using molecular assays.
Growth of high grade prostate cancer (e.g. Gleason grade 4/5) | following 2-6 weeks of cholesterol lowering intervention.
  Prostate tissue removed at the time of surgery will be examined to measure cellular growth using molecular assays.

CONTACTS AND LOCATIONS:
Overall Officials: Hyung L Kim, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States